CLINICAL TRIAL: NCT06573125
Title: Feasibility and Preliminary Efficacy of an App-Based Physical Activity Intervention for Individuals With Depression (MoodMover): A Protocol for a Single-Arm, Pre-Post Intervention Study
Brief Title: A Feasibility and Preliminary Efficacy Study of an App-Based Physical Activity Intervention (MoodMover) for Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Guy Faulkner, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H24-01820
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Depression
Keywords: mHealth; Physical Activity; Behavior Change; Mental Health; eHealth
MeSH Terms: conditions — Depression; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single-Arm, Pre-Post Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MoodMover (Experimental): Participants engage with MoodMover regularly as instructed over a period of 9 weeks, along with a 9-week follow-up.
  Interventions: Behavioral: MoodMover

INTERVENTIONS:
Behavioral: MoodMover — MoodMover is a 9-week app-based program aimed at increasing physical activity (PA) among individuals with depression, delivered via Pathverse. The current version of MoodMover includes one introductory module for baseline self-monitoring, eight primary modules, and eight optional supplementary modules. The program uses a variety of formats to deliver educational content, including videos, podcasts, and illustrated articles. In addition to its structured psychoeducational content, the app provides a range of behavioral features.

SUMMARY:
Exercise is recommended as a standalone treatment for mild-to-moderate depression in Canada. However, it's unclear how mental health practitioners can guide patients to structured, in-person exercise programs. In cases where such programs are not available or are unattractive to some, self-guided mobile health physical activity interventions could be a potential alternative. The investigators have been following a behavioural intervention development framework to create a 9-week, app-based physical activity intervention called MoodMover for people with depression. To evaluate the feasibility and preliminary efficacy of MoodMover, this study will employ a single-arm, pre-post experimental trial.

DETAILED DESCRIPTION:
MoodMover is a 9-week, app-based physical activity intervention, comprising a one-week run-in period, followed by eight major lessons, each complemented by an optional lesson, with new lessons becoming available on a weekly basis. Each major lesson addresses a specific topic designed to enhance physical activity engagement, covering topics including 1) feeling better through daily activity, 2) making physical activity enjoyable, 3) building self-confidence, 4) building physical activity opportunities, 5) developing self-regulatory skills, 6) drawing on social support, 7) forming an exercise habit, and 8) building exercise identity. Key features include step tracker, exercise logging with mood monitoring, action planning, gamification, and anonymized communications among users.

PRIMARY OBJECTIVE: This trial primarily aims to evaluate the feasibility and acceptability of MoodMover. In addition, the study will preliminarily assess the efficacy of MoodMover by monitoring changes in daily step counts, the main behavioral outcome of interest. Furthermore, the study will assess alterations in depressive symptoms and explore the association between these changes.

RESEARCH METHODOLOGY: All participants will begin by completing baseline assessments on REDCap. They will then participate in a 15-minute orientation session via Zoom with a researcher on the program's start date. The first five orientation sessions will be recorded and evaluated by an independent researcher using a fidelity checklist, allowing for immediate improvements in treatment fidelity. Following the orientation, participants will use MoodMover as directed for the duration of the 9-week program. No additional support will be offered except for technical issues. After completing the intervention, participants will undergo a follow-up assessment on REDCap. Participants will be encouraged to keep the app on their smartphones and continue using it after the program concludes. If they choose not to uninstall the app, this will be considered implied consent for the researcher to monitor their ongoing user engagement and physical activity data for an additional 9-week follow-up period. At the end of this period, participants will be contacted to sync their step data with MoodMover, enabling the collection of physical activity data throughout the follow-up. Additionally, participants will be asked to complete a satisfaction survey on REDCap.

STATISTICAL ANALYSIS: The analysis will involve (1) Descriptive statistics, (2) Regression-based analyses to evaluate the relationships between feasibility outcomes and other variables, and (3) Random effects mixed modeling to assess the impact of MoodMover on secondary outcomes and the relationship between changes in physical activity and depressive symptoms. As an underpowered single-arm feasibility study, the reporting of efficacy outcomes will focus on estimation.

ELIGIBILITY:
Inclusion Criteria:

AGE: 18-64 years DIAGNOSIS: A self-reported current diagnosis of major depressive disorder and/or at least mild depressive symptoms (>= 5) on the Patient Health Questionnaire, 9-Item (PHQ-9).

DEVICE: Possess an iPhone or Android smartphone with internet access to download the app.

LANGUAGE: Read, write understand, and communicate in the English language (or as appropriate)

Exclusion Criteria:

1. Are experiencing acute risk of harm to self or others
2. Have an active alcohol or substance use disorder
3. Physical disability preventing exercise
4. Active psychosis or mania
5. Severe cognitive impairment
6. Current pregnancy
7. Patients whose depression is directly linked to another major primary psychiatric disorder, such as psychosis or bipolar disorder
8. Exercise >= 90 min moderate-vigorous physical activity per week or >= 3 times/week
9. Anticipate a major absence (e.g., long vacation, surgery) in the next 3 months
10. Anticipate a major change to participants' current antidepressant treatment regimen (if any, e.g., medications, psychotherapy) in the next 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate assessed by the proportion of enrolled participants to those who are eligible and interested. | After recruitment is completed (up to 6 months)
  Successful recruitment will be defined as achieving a rate of 65%.
Intervention adherence assessed by the proportion of participants who complete the majority of major lessons. | Post-intervention (week 10)
  An adherence rate of 70% will be deemed as acceptable.
User Engagement: Time spent on each module will be downloaded from the Pathverse admin web portal. | Post-intervention (week 10) and up to 18 weeks
  Time spent on each module will be generated by Pathverse and reported in seconds.
Usability assessed by the adapted, patient version of the mHealth app usability questionnaire (MAUQ) for standalone apps. | Post-intervention (week 10)
  An average score of 5 and over will be deemed as acceptable.
Retention rates indicated by the proportion of participants completing both pre- and post-intervention questionnaires. | Post-intervention (week 10)
  An attrition rate of 30% will be defined as acceptable.
Compliance to the graded goal setting indicated by the proportion of participants who successfully set their step goals as instructed. | During the intervention (weeks 2-9) and Post-intervention (week 10)
  The proportion of participants who successfully set their step goal in week 2, and those who modified their step goals in week 4 and week 6, will be reported separately. Participants who followed all the instructions across these time points will be deemed as having achieved "full compliance", while those who followed instructions at one or two time points will be deemed as having achieved "partial compliance". Participants who did not follow instructions at any time points will be deemed as having achieved "no compliance".
User satisfaction assessed by Melin et al.'s mHealth Satisfaction Questionnaire (14-item) | Post-intervention (week 10) and 9-week follow-up (week 18)
  Melin et al.'s mHealth Satisfaction Questionnaire is a 14-item questionnaire. Scores range from 0 to 60, with higher scores indicating better satisfaction levels.

SECONDARY OUTCOMES:
Device-based physical activity assessed by the smartphone's built-in step counting function | Baseline (week 1), during the intervention (weeks 1- 9), post-intervention (week 10), and follow-up (week 18)
  Daily step counts will be collected using the smartphone's built-in step counting function.
Subjective physical activity assessed by the Canadian Physical Activity Adult Questionnaire (PAAQ) | Enrollment (week 0) and post-intervention (week 10)
  This questionnaire is designed in accordance with the Canadian Physical Activity Guidelines, which recommend a minimum of 150 minutes of MVPA per week for adults. It has been widely employed for monitoring PA in Canadian adults.
Depressive symptoms assessed by the Patient Health Questionnaire-9 (PHQ-9) | Enrollment (week 0) and post-intervention (week 10)
  The Patient Health Questionnaire-9 (PHQ-9) is a validated, self-administered tool for assessing depression. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Anxiety assessed by the Generalized Anxiety Disorder 7 scale (GAD-7) | Enrollment (week 0) and post-intervention (week 10)
  The Generalized Anxiety Disorder 7 scale (GAD-7) is a seven-item validated instrument for measuring the severity of anxiety. Scores range from 0 to 21, with higher scores indicating more severe anxiety.
Sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI) | Enrollment (week 0) and post-intervention (week 10)
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated, 19-item questionnaire that assess sleep-related problems. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Functional disability assessed by the short-version of the World Health Organization Disability Assessment Schedule 2.0 | Enrollment (week 0) and post-intervention (week 10)
  The short-version of the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) will be utilized. Scores range from 0 to 100, with higher scores indicating more severe disability.
Affective attitudes assessed using items derived from Tang et al. (2023) | Enrollment (week 0) and post-intervention (week 10)
  Affective attitudes will be measured on three 7-point bipolar scales (Unenjoyable (1) to enjoyable (7); Boring (1) to very exciting (7); Unpleasant (1) to very pleasant (7)). All items share the same stem: "For me, participating in regular PA over the next month would be ..." Higher scores indicate more positive attitudes.
Instrumental attitudes assessed using items derived from Tang et al. (2023) | Enrollment (week 0) and post-intervention (week 10)
  Instrumental attitudes will be measured on three 7-point bipolar scales (Unwise (1) to very wise (7); Not beneficial (1) to very beneficial (7); Useless (1) to very useful (7)). All items share the same stem: "For me, participating in regular PA over the next month would be ..." Higher scores indicate more positive attitudes.
Perceived opportunity assessed using items derived from Tang et al. (2023) | Enrollment (week 0) and post-intervention (week 10)
  Perceived opportunity will be assessed using three 5-point Likert scales, ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher perceived opportunity.
Perceived capability assessed using items derived from Tang et al. (2023) | Enrollment (week 0) and post-intervention (week 10)
  Perceived capability will be assessed using three 5-point Likert scales, ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher perceived capability.
Intention strength assessed using items derived from Tang et al. (2023) | Enrollment (week 0) and post-intervention (week 10)
  Intention strength will be measured using three items (e.g., I am committed to engage in physical activity over the next month). Participants will rate these items on 5-point Likert scales ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher intention strength.
Decisional intention assessed using item "I intend to increase 3000 steps above my baseline daily steps for most days per week." | Enrollment (week 0) and post-intervention (week 10)
  Participants will be asked to provide binary responses (Yes/No).
Regulations assessed using items derived from Rovniak et al. 2002. | Enrollment (week 0) and post-intervention (week 10)
  Regulations will be measured using 5-point Likert scales with three items pertaining to self-monitoring, goal-setting, and action planning. Higher scores indicate stronger regulatory skills.
Habit assessed using items modified from Rhodes and Lim (2016) | Enrollment (week 0) and post-intervention (week 10)
  Habit will be assessed using 5-point Likert scales with three items (e.g., "I engage in regular physical activity without having to consciously remember it"). Higher scores indicate stronger habit.
Identity assessed using items modified from Rhodes and Lim (2016) | Enrollment (week 0) and post-intervention (week 10)
  Identity will be measured using 5-point Likert scales with three items (e.g., "When I describe myself to others, I usually include my involvement in physical activity"). Higher scores indicate a stronger exercise identity.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Faulkner, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang Y, Gierc M, La H, Kim J, Liu S, Lam RW, Puterman E, Faulkner G. MoodMover: Development and usability testing of an mHealth physical activity intervention for depression. Digit Health. 2025 Feb 3;11:20552076251317756. doi: 10.1177/20552076251317756. eCollection 2025 Jan-Dec. PMID 39906877
- [Background] Rhodes RE, Lim C. Understanding action control of daily walking behavior among dog owners: a community survey. BMC Public Health. 2016 Nov 16;16(1):1165. doi: 10.1186/s12889-016-3814-2. PMID 27852251
- [Background] Tang Y, Gierc M, Whiteford V, Rhodes RE, Faulkner G. Exploring correlates of physical activity using the multi-process action control framework: is there a moderating role for mental health? International Journal of Sport and Exercise Psychology. 2023:1-19. doi: https://doi.org/10.1080/1612197X.2023.2225515.
- [Background] Rovniak LS, Anderson ES, Winett RA, Stephens RS. Social cognitive determinants of physical activity in young adults: a prospective structural equation analysis. Ann Behav Med. 2002 Spring;24(2):149-56. doi: 10.1207/S15324796ABM2402_12. PMID 12054320
- [Derived] Tang Y, Gierc M, La H, Liu S, Lam RW, Puterman E, Faulkner G. Feasibility and preliminary effects of an app-based physical activity intervention for individuals with depression (MoodMover): A protocol for a single-arm, pre-post intervention study. PLoS One. 2025 Apr 22;20(4):e0321958. doi: 10.1371/journal.pone.0321958. eCollection 2025. PMID 40261856